CLINICAL TRIAL: NCT01156181
Title: Effect of Cervical Discharge Removal Before Embryo Transfer on ICSI Cycle Outcomes
Brief Title: Effect of Cervical Discharge Removal During ET on Pregnancy Rate
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Emb-007
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2010-07

CONDITIONS: Infertility
Keywords: Cervical mucus, Embryo transfer, ICSI cycle, Pregnancy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical discharge removal (Experimental): Cervical discharge will be removed using a cotton swab before embryo transfer during ICSI cycles
  Interventions: Procedure: Cervical discharge removal
- Control (Active Comparator): Embryo transfer without any intervention
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: Cervical discharge removal — Cervical discharge will be removed using a cotton swab before embryo transfer during ICSI cycles
  Arms: Cervical discharge removal
Procedure: control — Embryo transfer without any intervention
  Arms: Control

SUMMARY:
Pregnancy rate may be affected by multiple factors such as embryo transfer techniques. Even small differences in embryo transfer methods may affect pregnancy rates. There is an inconsistency about the effect of the removal of cervical discharge on embryo transfer outcomes. Some studies showed that cervical mucus removal before embryo transfer can increase pregnancy rate, however the others could not find any significant effect about the removal of cervical mucus on pregnancy or live birth rates. Given to the conflicting evidences, our study aimed to determine whether the cervical discharge removal has positive effect on pregnancy rate.

DETAILED DESCRIPTION:
492 Infertile women who were candidate for fresh embryo transfer during IVF/ICSI cycles were eligible for this study if they had two or more good quality embryos. All categories of female or male factors infertility except uterine factor infertility were eligible for participation in the study. Immediately prior to embryo transfer, women were randomly allocated to either treatment (cleaning the cervical canal) or control groups. In treatment group, excess mucus and debris were cleared from the cervical canal using a sterile cotton swabs. The cervical discharge was scored as mucosal, bloody, combination of mucosal and bloody, or infected. Control group had no cervical cleaning before embryo transfer. Then, the embryos were loaded into the transfer catheter by the embryologist and were deposited into the uterine cavity by one experience physician. The primary endpoint was clinical pregnancy. Fertilization, Implantation, abortion, and live birth rates were the other outcomes of interest or secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who were candidate for fresh embryo transfer during IVF/ICSI cycles were eligible for this study if they had two or more good quality embryos and age fewer than 40

Exclusion Criteria:

* The patients with frozen-thawed embryo transfer cycle
* Those with oocyte donation cycle
* The women with uterine abnormality
* The women with submucosal and intramural myoma
* Who does not have good-quality embryos appropriate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 492 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 9 months after recruiting

SECONDARY OUTCOMES:
Fertilization rate | 2 weeks
Implantation rate | 1 month
Miscarriage rate | 9 months
Live birth rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Moini Moini, MD, Study Chair — Academic staff of Endocrinology and Female Infertility Department, Royan Institute, Tehran - Iran; Ladan Mohammadi yeganeh, MSc, Principal Investigator — Investigator
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Moini A, Kiani K, Bahmanabadi A, Akhoond M, Akhlaghi A. Improvement in pregnancy rate by removal of cervical discharge prior to embryo transfer in ICSI cycles: a randomised clinical trial. Aust N Z J Obstet Gynaecol. 2011 Aug;51(4):315-20. doi: 10.1111/j.1479-828X.2011.01318.x. Epub 2011 Jun 9. PMID 21806579
- See also: Related Info — http://www.royaninstitute.org